CLINICAL TRIAL: NCT05568914
Title: Intra Dialytic Parenteral Nutrition During Intermittent Hemodialysis Can Close the Nutritional Gap Identified by Indirect Calorimetry: a Pilot and Feasibility Study
Brief Title: Intra Dialytic Parenteral Nutrition and Nutritional Gap Nutritional Gap Identified by Indirect Calorimetry
Acronym: DiaPaNIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-EDW-DiaPaNIC
Record Dates: First submitted 2022-08-30; First posted 2022-10-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Chronic Kidney Diseases; Protein Energy Wasting
Keywords: Indirect Calorimetry; Parenteral Nutrition; Hemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphagia | interventions — Calorimetry, Indirect; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assessments (Experimental): In this single-arm trial, each participant undergoes the following measurements/assessments:
  Physical: Body weight (before and after dialysis), length Biophysical: NRS2002, GLIM, Bio-electrical Impedance Analysis Metabolic: Indirect Calorimetry Nutritional: dietary anamnesis, 3-days nutritional diary
  Interventions: Device: Indirect Calorimetry; Device: Bio-electrical Impedance Analysis (BIA); Other: Nutritional assessments

INTERVENTIONS:
Device: Indirect Calorimetry — Indirect Calorimetry (Q-NRG Metabolic Monitor, COSMED) is performed to determine the Resting Energy Expenditure before hemodialysis.
  Other Names: Q-NRG Metabolic Monitor, COSMED
Device: Bio-electrical Impedance Analysis (BIA) — Bio-electrical Impedance Analysis (BIA101/BIVA, Akern) is used to analyse the body composition (Fat Mass, Fat Free Mass, Phase Angle).
  Other Names: BIA101/BIVA, Akern
Other: Nutritional assessments — The Nutritional assessments consist of a dietary anamnesis and a 3-day nutritional diary to determine the nutritional (caloric and protein) intake of the participants.
  Other Names: Dietary anamnesis; Nutritional diary

SUMMARY:
Renal failure is a relevant condition as the incidence of patients treated with intermittent dialysis continues to grow each year. One of the strongest predictors of mortality in these patients is Protein-Energy Wasting (PEW). Optimal nutritional support, combined with physical exercise may be able to improve the physical condition objectified as muscle wasting and weakness. Correct nutritional support must aim to supplement the correct combination of protein and caloric needs. Although no other way exist than predicting formula to assess protein need, predicting formula don't seem to capture the individual caloric need of the patients. The gold standard to assess caloric need by measuring Resting Energy Expenditure (REE) is indirect calorimetry. Even when caloric and protein targets are defined, intake remains a challenge because of intake restriction in dietary patterns. This is why intradialytic parenteral nutrition (IDPN) can play an crucial role for closing the nutritional gap. Whether IDPN guided by indirect calorimetric measurements of metabolism can close the gap when oral intake fails, remains an unanswered question.

DETAILED DESCRIPTION:
Renal failure is a relevant condition as the incidence of patients treated with renal replacement therapy and specifically intermittent dialysis, continues to grow each year. In 2021 up to 4845 patients required intermittent dialysis in Flanders, Belgium. Weight loss and homeostatic disturbances of energy and protein balances are often present in Chronic Kidney disease (CKD) and end-stage renal disease (ESRD).The international society of renal nutrition and metabolism defines Protein-Energy Wasting (PEW) as the state of nutritional and metabolic disorders in patients with CKD and ESRD, characterized by simultaneous loss of systemic body protein and energy stores. PEW is one of the strongest predictors of mortality in CKD patients. Up tot 54% of adults undergoing chronic intermittent haemodialysis (IHD) suffer from PEW due to a combination of the disease and therapy. Adequate nutritional therapy can reverse the negative impact of PEW. Optimal nutritional support, next to physical exercise may be able to improve the physical condition objectified as muscle wasting and weakness. Correct nutritional support must aim to supplement the correct combination of protein and caloric after assessing the needs and intake of different nutrients. Although no other way exist than predicting formula to assess protein need, predicting formula don't seem to capture the individual caloric need of the patients. The gold standard to assess caloric need by measuring Resting Energy Expenditure (REE) is indirect calorimetry. This technique measures the individual VCO2 and VO2 and after integrating it into the Weir equation it calculates REE. Even when caloric and protein target are defined, intake remains a challenge because of intake restriction in dietary patterns. This is why intradialytic parenteral nutrition (IDPN) can play an crucial role for closing the nutritional gap. In clinical practice, in 38% of dialysis patients, IDPN is used. The most common IDPN were triple phase bags. Whether IDPN guided by indirect calorimetric measurements of metabolism can close the gap when oral intake fails, remains an unanswered question.

ELIGIBILITY:
Inclusion Criteria:

* Patient on intermittent hemodialysis
* Protein-Energy Wasting defined as 5% within 3 months or 10% within 6 months (not due to water loss, established at the discretion of the treating physician)

Exclusion Criteria:

* Pregnancy
* Contra-indications for the use of indirect calorimetry as stated by the AARC (oxygen therapy for COPD,...)
* Metabolic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Caloric adequacy | Pre-dialysis
  caloric intake (kcal/day) and caloric need (kcal/day) (see secondary outcomes) will be combined to report caloric adequacy according to this equation: [sum of percentage of caloric intake/caloric need]/total of evaluable nutrition days (%)

SECONDARY OUTCOMES:
Protein adequacy | Pre-dialysis
  protein intake (from nutritional assessments)/protein need (%)
Fat Mass (FM) | 20-30 minutes after dialysis
  measured by Bio-electrical Impedance Analysis (BIA) (kg and %);
Fat Free Mass (FFM) | 20-30 minutes after dialysis
  measured by Bio-electrical Impedance Analysis (BIA) (kg and %);
Phase angle | 20-30 minutes after dialysis
  measured by Bio-electrical Impedance Analysis (BIA) (kg and %);
Body weight | before and after hemodialysis
  Body weight (kg)
Compatibility between the caloric gap and PN ready to use formulae on the market | through study completion or one year, whichever is sooner
  Comparison between individual caloric need of patients and ready to use PN formulae (PeriOlimel N4E (Baxter), Olimel N5E (Baxter), Olimel N7E (Baxter), Olimel N9/N9E (Baxter), Olimel N12/N12E (Baxter), SMOFKabiven Ex-tra Amino (Fresenius), SMOFKabiven peripheral (Fresenius), SMOFKabiven Peri Low Osmo (Fresenius), SMOFKabiven E/EF (Frese-nius), Omegomel Peri (Baxter), Nutriflex Omega Special (B Braun); based on caloric content per bag of PN on the market (Unit of measurement: portion of PN bag (%) needed to close the caloric gap)
Mean caloric intake | pre-dialysis
  (kcal/day) from nutritional assessments (3-day nutritional diary and nutritional anamnesis
Caloric need | pre-dialysis
  (kcal/day): Resting Energy Expenditure (REE) measured by Indirect Calorimetry (IC)
Mean protein intake | pre-dialysis
  g/day): from nutritional assessments (3-day nutritional diary and nutritional anamnesis
Barriers for patients for use of IDPN | pre-dialysis
  "would you agree to IDPN if your health condition required it? Please elaborate"
Barriers for dialysis nurses and nephrologists for use of IDPN | throughout the duration of the trial
  "Are logistical and practical barriers holding you back from prescribing or administering IDPV? Please elaborate."

OTHER OUTCOMES:
Descriptive outcomes | pre-dialysis
  age, sex, category of kidney disease, comorbidities, dialysis vintage (years)
Dialysis type | During dialysis
  (from medical file)
Delta REE between predicting formula and indirect calorimetry | Pre-dialysis
  Difference in energy need as calculated using standard formula and measured using IC
Vascular access type | during dialysis
  (from medical file)
Dialysis blood flow rate | During dialysis
  (from medical file)
Hemodialysis treatment adequacy (kt/V) | During dialysis
  (from medical file)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth De Waele, MD, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No